CLINICAL TRIAL: NCT06051071
Title: Home-based Transcranial Direct Current Stimulation to Modulate Neural Networks and Promote Resilience
Brief Title: Home-based Stimulation to Promote Resilience
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Guttmann (Other)
Collaborators: University of Barcelona (Other)
Responsible Party: Principal Investigator, Javier Solana Sanchez, Principal Investigator, Institut Guttmann
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201129-30-31
Record Dates: First submitted 2023-06-30; First posted 2023-09-22 (Actual); Last update posted 2023-09-22 (Actual); Status verified 2023-09

CONDITIONS: Stress
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): tDCS stimulation arm
  Interventions: Device: Transcranial Direct Current Stimulation (tDCS)

INTERVENTIONS:
Device: Transcranial Direct Current Stimulation (tDCS) — In tDCS, surface electrodes (anode and cathode) inject low-intensity direct current through the skull to modulate brain activity and cortical excitability

SUMMARY:
Background:

Non-invasive brain stimulation showed to be effective in reduce stress related cognitive and mental-health consequences. Thanks to technological advances these devices are now very easy to use and suitable to hoe-based self-administration.

Objective:

Conduct a home-based and tele-supervised non-invasive brain stimulation intervention to modulate the expression of resilience brain networks.

Methods:

Transcranial direct current stimulation will be used duringa tele-supervised home-based stimulation intervention to promote the expression of brain resilience networks.

Expected results:

The present project should provide critical new knowledge and evidences of the feasibility and impact of modulating brain resilience networks in terms of its effects on mental health of participants, including the possibility to implement future self-administered, home-based interventions.

DETAILED DESCRIPTION:
Resilience, the concept that describes the ability of certain individuals to resist, among others, the impact of stress, is a broad term.

In clinical psychology and mental health, the concept of resilience has historically been linked to the study of individual differences (e.g. self-esteem, sense of control, perception of social support, etc.) that determine the ability to cope with the impact of life traumas and maintain good psychological and physical functioning, avoiding mental illness.

Neuroimaging research has identified brain regions that show patterns of specific activity and connectivity during exposure to stressful or violent stimuli and may be correlated with scores on psychosocial resilience scales or predict coping capabilities.

In the same vein, our group has recently observed how certain connectivity patterns between frontal and parietal areas related to the default neural network (DMN) and pedimental-parietal network (FPN), are predictive of better stress resilience, which decreases the negative impact on mental health.

Together, these findings suggest the possible existence of brain circuits composed of nodes within medial dorsolateral and prefrontal brain areas, and their connections to parietal areas, specifically related to resilience capacity.

In this context non-invasive transcranial stimulation, a safe and effective procedure, provides us with a technique to modulate brain activity in these areas and potentially promote resilience.

Among the various techniques, direct current transcranial stimulation (tDCS) is one of the most studied and promising approaches.

In tDCS, surface electrodes (anode and cathode) inject low-intensity direct current through the skull to modulate brain activity and cortical excitability, with regulatory effects affecting not only areas brains stimulated, but also connected brain networks, and thus with the potential to "optimize" the balance between integration and segregation of associated functions.

Crucially, advances in technology have made tDCS devices more portable and user-friendly, with the possibility of being configured at a distance, and potentially allowing their home administration, with remote supervision, facilitating adherence to intervention protocols.

Goal The aim of this study is to assess the feasibility and effects of a direct intervention to promote resilience to stress

Materials and Method Study Design The researchers will implement an open trial with healthy adults performing a pre-stimulation assessment, a remotely supervised home intervention with tDCS, and a post-treatment assessment.

During the previous assessment, participants will receive training on the use of the stimulation device, as well as information material, and over the course of the intervention, and for the duration of the intervention researchers will remotely monitor the stimulation.

Participants This study will involve 40 healthy adults aged 40 to 65. The sample size has been calculated taking into account the grandor effect of previous studies investigating the modulating effect of non-invasive brain stimulation on functional and behavioral aspects related to resilience, defined as the ability to resist external and stressful factors.

The size of the required sample, considering alpha=0.05 and statistical power (1-beta) =0.80, has been estimated at between 30 and 38 individuals depending on the statistical test. Considering a possible abandonment of around 10%, the final sample will consist of 40 individuals.

Pre-Post Assessment Prior to the intervention, participants will be administered with questionnaires and a paradigm of stress induction.

Once the intervention is complete, the same tests will be repeated.

Stress Induction Paradigm In this task, developed by Limbachia and collaborators there are two circles that move at times by approaching and sometimes moving away from each other. When the circles are touched, the participants receive a soft electrical stressor stimulus. Circular motion has a high degree of unpredictability.

The stressful electric stimulus will be delivered by 500 ms through electrodes, to the fourth and fifth fingers of the left hand. To gauge the intensity of the shock, each participant will be asked to choose their own level of stimulation before the stress task, so that the stimulus is "unpleasant but not painful".

During the task, changes in skin conduction, heart rate, pupil diameter and changes in connectivity and network oscillation reflected by the signal electroencephalography will be recorded.

Feasibility Indicators To confirm the feasibility of such interventions, the investigators will evaluate adherence to intervention.

Stimulation training the researchers will undertake a first training session in person, followed by a training and remote monitoring program. These training sessions will aim to instruct and ensure the correct administration of stimulation.

Stimulation sessions oversight

The researchers will carry out remote monitoring throughout the duration of the intervention:

Investigators will monitor the first 2/3 stimulation sessions, second needs, and until participants need it. From the second week on, researchers will follow the intervention weekly through at least one video call per week.

TDCS stimulation protocol:

The stimulation session will last 20 minutes, following a protocol widely used in various studies.

Stimulation will be performed in the left dorsal lateral prefrontal cortex (L-DLPFC).

The current will be supplied steadily for 30 minutes and all the stimulation parameters to be used adhere to the general guidelines of the safety criteria of transcranial electric stimulation and, for safety reasons, the maximum supplied current will be 2 ma.

The stimulation will be delivered using the Sooma tDCSTM medical device used by health professionals worldwide. This device has acquired CE, Health Canada, MDA, HSA, TGA and COFEPRIS approvals. Sooma tDCSTM devices are manufactured in Finland under ISO 13485 standard.

ELIGIBILITY:
Inclusion Criteria:

* No psychiatric conditions or neurological disorders
* Do not present any contraindication for their safety in relation to the TDCS protocol (crew metal implants, pacemakers, medical infusion bomb, epilepsy history, brain surgeries, etc.)

Exclusion Criteria:

* alcohol or drug abuse
* pregnancy

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-15 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in the Connor Davidson resilience scale | immediately after the intervention
  A resilience scale scoring from 0 to 40, where higher score represent better resilience
Changes in the State-Trait Anxiety Inventory | immediately after the intervention
  Anxiety scale scoring from 0 to 80 where higher scores indicates greater anxiety
Changes in the Holmes stress inventory | immediately after the intervention
  stress scale scoring from 0 to 430 points, where higher scores indicates greater stress
Adherence | immediately after the intervention
  number of sessions completed

SECONDARY OUTCOMES:
Heart rate variability changes | immediately after the intervention
  Heart rate changes during the task
Pupill dilatation changes | immediately after the intervention
  Pupil diameter changes during the task
Skin electrical activity changes | immediately after the intervention
  Skin electrical activity changes during the task
EEG signal changes | immediately after the intervention
  EEG signal changes during the task

CONTACTS AND LOCATIONS:
Locations (1):
- Guttmann Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided